CLINICAL TRIAL: NCT05357560
Title: A Phase Ib Multi-stage Plasmodium Falciparum Malaria Vaccine Study to Assess the Safety and Immunogenicity of the Blood-stage Vaccine Candidate RH5.2 Virus-like Particle (VLP) in Matrix-M and the Pre-erythrocytic Stage Vaccine Candidate R21 in Matrix-M, Both Alone and in Combination, in Adults and Infants in the Gambia
Brief Title: A Study to Assess the Experimental Malaria Vaccines RH5.2-VLP and R21
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Medical Research Council Unit, The Gambia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC086
Record Dates: First submitted 2022-04-13; First posted 2022-05-03 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Malaria, Plasmodium Falciparum
Keywords: RH5.2 virus-like particle (VLP); Matrix-M; R21
MeSH Terms: conditions — Malaria, Falciparum | interventions — Matrix-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group 1 - Infants R21 delayed 3rd dose (Experimental): 11 volunteers (infant 5-17 months) given 50 µg of Matrix-M in combination with 5µg R21 at months 0, 1 and 6 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 2 - Infants R21 standard regimen (Experimental): 11 volunteers (infant 5-17 months) given 50 µg of Matrix-M in combination with 5µg R21 at months 0, 1 and 2 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 3 - Adults RH5.2 low dose, standard regimen (Experimental): 10 volunteers (adult 18-45 years) given 50 µg of Matrix-M in combination with 10µg RH5.2 VLP at months 0, 1 and 2 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 4 - Adults RH5.2 high dose, standard regimen (Experimental): 10 volunteers (adult 18-45 years) given 50 µg of Matrix-M in combination with 50µg RH5.2 VLP at months 0, 1 and 2 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 5 - Adults RH5.2 and R21 low dose, standard regimen (Experimental): 10 volunteers (adult 18-45 years) given 50 µg of Matrix-M in combination with 10µg RH5.2 VLP and 10µg R21 at months 0, 1 and 2 via intramuscular (IM) injection in the deltoid region of the non-dominant arm
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 6 - Infants RH5.2 standard regimen (Experimental): 11 volunteers (infant 5-17 months) given 50µg of Matrix-M in combination with 5µg RH5.2 VLP at months 0, 1 and 2 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 7 - Infants RH5.2, delayed 3rd dose (Experimental): 11 volunteers (infant 5-17 months) given 50µg of Matrix-M in combination with 5µg RH5.2 VLP at months 0, 1 and 6 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 8 - Infants RH5.2 and R21, standard regimen (Experimental): 11 volunteers (infant 5-17 months) given 50µg of Matrix-M in combination with 5µg RH5.2 VLP and 5µg R21 at months 0, 1 and 2 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21
- Group 9 - Infants RH5.2 and R21, delayed 3rd dose (Experimental): 11 volunteers (infant 5-17 months) given 50µg of Matrix-M in combination with 5µg RH5.2 VLP and 5µg R21 at months 0, 1 and 6 via intramuscular (IM) injection in the anterolateral thigh
  Interventions: Biological: Matrix-M with RH5.2 VLP and/or R21

INTERVENTIONS:
Biological: Matrix-M with RH5.2 VLP and/or R21 — 3 doses of 50 µg of Matrix-M in combination with RH5.2 VLP and/or R21 at different doses and at different timepoints

SUMMARY:
This is a Phase Ib multi-stage Plasmodium falciparum malaria vaccine study to assess the safety and immunogenicity of the blood-stage vaccine candidate RH5.2 virus-like particle (VLP) in Matrix-MTM and the pre-erythrocytic stage vaccine candidate R21 in Matrix-MTM, both alone and in combination, in adults and infants in the Gambia

DETAILED DESCRIPTION:
A total of 96 volunteers will be enrolled. Adults (18-45 years) will be enrolled into groups 3 -5. Infants (5 -17 months) will be enrolled into groups 1-2 and groups 6-9. All volunteers will be given 3 doses 50 µg of Matrix-M in combination with RH5.2 VLP and/or R21 via intramuscular (IM) injection in the deltoid region of the non-dominant arm for adults and anterolateral thigh for infants. The first 2 doses will be given at months 0 and 1. Groups 2-6 and group 8 will be given the third dose at month 2, and groups 1, 7 and 9 will be given the third dose at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1, 2 and 6-9: Healthy male or female infants aged 5-17 months at the time of enrolment with signed consent obtained from parents or guardians.
* Groups 3-5: Healthy male or female adults aged 18-45 years at the time of enrolment with signed consent.
* Groups 3-5 (Female participants only): Must be non-pregnant (as demonstrated by a negative urine pregnancy test), and practice continuous effective contraception for the 24 to 30 month duration of the study (see section 9.9).
* Planned long-term (at least 24 months from the date of recruitment) or permanent residence in the study area.
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or infants with Z-score of weight-for-age within ±2SD.

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual
* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease and neurological illness as judged by the PI or other delegated individual.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g., Kathon, neomycin, betapropiolactone.
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality at grade 2 or above as judged by the PI or other delegated individual.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination. This excludes COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination, and EPI vaccines (for infants), which should not be received between 14 days before to 28 days after any study vaccination.
* History of vaccination with previous malaria vaccines
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment in adults or at any time for infants, or planned use during the study period.
* Suspected or known current alcohol abuse.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV IgG) or HIV. For infants, any history of vertical exposure to HIV infection.
* Any other finding which in the opinion of the PI or other delegated individual would increase the risk of an adverse outcome from participation in the trial.
* Positive malaria by PCR screening.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Vaccination and re-vaccination exclusion criteria

The following events associated with vaccine immunisation constitute absolute contraindications to further administration of vaccine. If any of these events occur during the study, the participant must be withdrawn and followed until resolution of the event, as with any adverse event:

* Anaphylactic reaction following administration of vaccine.
* Pregnancy. The following adverse events constitute contraindications to administration of vaccine at that point in time; if any one of these adverse events occurs at the time scheduled for vaccination, the participant may be vaccinated at a later date, or withdrawn at the discretion of the Investigator.

The participant must be followed until resolution of the event as with any adverse event:

* Acute disease at the time of administration of the IP (acute disease is defined as the presence of a moderate or severe illness with or without fever or symptoms suggestive of possible COVID-19 disease). All vaccines can be administered to persons with a minor illness such as diarrhoea or mild upper respiratory infection without fever, i.e. axillary temperature < 37.5°C.
* Temperature of >37.5°C (99.5°F) at the time of vaccination.
* Confirmed current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR swab or rapid antigen test taken during current illness or positive COVID-19 PCR swab or rapid antigen test within preceding 7 days without symptoms. Vaccinations will be delayed by a minimum of 7 days from the date of the first positive COVID-19 PCR swab, as long as symptoms are improving or resolved and there is no fever. It will be at the discretion of the Investigator to withdraw a participant if they develop severe COVID-19 disease.

Ages: 5 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To determine safety and tolerability of RH5.2-VLP with Matrix-M and R21 with Matrix-M, in healthy adults and infants by assessing the occurrence of solicited local reactogenicity signs and symptoms via clinic and home visits | 7 days following each vaccination
  Occurrence of solicited local reactogenicity signs and symptoms via clinic and home visits
To determine safety and tolerability of RH5.2-VLP with Matrix-M and R21 with Matrix-M, in healthy adults and infants by assessing the occurrence of solicited systemic reactogenicity signs and symptoms via clinic and home visits | 7 days following each vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms via clinic and home visits
To determine safety and tolerability of RH5.2-VLP with Matrix-M and R21 with Matrix-M, in healthy adults and infants by assessing occurrence of unsolicited adverse events | 28 days following the vaccination
  Occurrence of unsolicited adverse events via clinical review, clinical examination (including observations) and laboratory results
Safety of the RH5.2-VLP with Matrix-M and R21 with Matrix-M vaccine, assessed through the number of participants with abnormal laboratory test results | 28 days following the vaccination
  Occurrence of change from baseline laboratory test results
Assessment of safety and tolerability of RH5.2-VLP with Matrix-M and R21 with Matrix-M, in healthy adults and infants assessed through the number of participants with serious adverse events | Whole duration of the study (24-30 months following initial trial vaccination)
  Occurrence of serious adverse events including grading of causality

SECONDARY OUTCOMES:
To assess the humoral and cellular immunogenicity of RH5.2-VLP with Matrix-M as assessed by magnitude assessment at various timepoint | From a number of key timepoints, baseline up to day 912 (dependant on group)
  RH5 serology (participants vaccinated with RH5.2-VLP only), blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for magnitude assessment, late timepoints used to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP with Matrix-M as assessed by antibody kinetics at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  RH5 serology (participants vaccinated with RH5.2-VLP only), blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for antibody kinetics, late timepoints used to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP with Matrix-M, performing ELISA at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  RH5 serology (participants vaccinated with RH5.2-VLP only), blood samples taken at a number of key timepoints performing ELISA at specified timepoints
To assess the humoral and cellular immunogenicity of R21 with Matrix-M performing ELISA at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  R21 serology (participants vaccinated with R21 only), blood samples taken at a number of key timepoints performing ELISA at specified timepoints
To assess the humoral and cellular immunogenicity of R21 with Matrix-M as assessed by antibody kinetics at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  R21 serology (participants vaccinated with R21 only), blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for antibody kinetics, late timepoints used to assess longevity of response
To assess the humoral and cellular immunogenicity of R21 with Matrix-M as assessed by magnitude assessment at various timepoint | From a number of key timepoints, baseline up to day 912 (dependant on group)
  R21 serology (participants vaccinated with R21 only), blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for magnitude assessment, late timepoints used to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M as assessed by antibody kinetics at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Hepatitis B serology, blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for antibody kinetics, late timepoints used to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M as assessed by magnitude assessment at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Hepatitis B serology, blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for magnitude assessment, and late timepoints to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M, performing ELISA at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Hepatitis B serology, blood samples taken at a number of key timepoints performing ELISA at specified timepoints
To assess the humoral and cellular immunogenicity of RH5.2-VLP with Matrix-M when administered to healthy volunteers at different doses and combinations and used in various regimens | Likely at V3+14 or V3+28
  Growth Inhibition Activity (GIA) (participants vaccinated with RH5.2-VLP only) performed at peak of response after the third vaccination, based on previous work this is likely to be at V3+14 or V3+28
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M as assessed by antibody kinetics at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Serum total IgG concentration determination, blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for antibody kinetics, late timepoints to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M as assessed by magnitude assessment at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Serum total IgG concentration determination, blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for magnitude assessment, late timepoints to assess longevity of response
To assess the humoral and cellular immunogenicity of RH5.2-VLP and R21 with Matrix-M, performing ELISA at various timepoints | From a number of key timepoints, baseline up to day 912 (dependant on group)
  Serum total IgG concentration determination, blood samples taken at a number of key timepoints performing ELISA at specified timepoints
To assess the humoral and cellular immunogenicity of R21 with Matrix-M when administered to healthy volunteers at different doses and combinations and used in various regimens | From a number of key timepoints, base line up to day 912 (dependant on group)
  Inhibition of sporozoite invasion assay (ISI) (participants vaccinated with R21 only), blood samples taken at a number of key timepoints including baseline and post vaccination of V+7 (adults only), V+14, V+28 to allow for antibody kinetics and magnitude assessment, and late timepoints to assess longevity of response, performing ELISA at every timepoint where 'immunology serum' is required

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Research Council Unit, Fajara, Banjul, The Gambia

REFERENCES:
- [Derived] Mo AX, McGugan G, Pesce JT. Meeting report: Expert consultation on late arresting replication competent (LARC) malaria sporozoite vaccine research & development. Vaccine. 2025 Apr 30;54:127009. doi: 10.1016/j.vaccine.2025.127009. Epub 2025 Apr 16. PMID 40245769